CLINICAL TRIAL: NCT06542965
Title: Clinical Characteristics, Risk Factors and Resistance Mechanisms for Bloodstream Infection of Carbapenem-Resistant Proteus Mirabilis
Brief Title: Bloodstream Infection of Carbapenem-Resistant Proteus Mirabilis
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Cağlar Iirmak, Principal Investigator, Medical Specialists in Infectious Diseases, Dokuz Eylul University
Other Study IDs: DEU-INF-IRMAK-1
Record Dates: First submitted 2024-07-31; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Proteus Mirabilis Infection; Bacteremia; Carbapenem Resistant Bacterial Infection
Keywords: Proteus mirabilis; bacteremia; carbapenem resistance; resistance mechanisms; PCR
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — blood culture samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case (Patients with carbapenem-resistant P. mirabilis): Patients with carbapenem-resistant P. mirabilis (CRPM) growth in blood culture were included in the case group
  Interventions: Other: Non-Interventional Research
- Control (Patients with carbapenem- susceptible P. mirabilis): Patients with carbapenem- susceptible P. mirabilis (CSPM) growth in blood culture were included in the control group
  Interventions: Other: Non-Interventional Research

INTERVENTIONS:
Other: Non-Interventional Research — Non-Interventional Research

SUMMARY:
This study aims to determine the clinical characteristics, risk factors, and resistance mechanisms of patients with carbapenem-resistant P. mirabilis bacteremia.Patients with P. mirabilis growth in blood culture samples sent to bacteriology laboratory between 2018 and 2021 were retrospectively analyzed. Patients meeting the inclusion criteria were divided into carbapenem-resistant and carbapenem- susceptible groups. The investigators recorded demographic data, clinical features, and laboratory findings. Resistance genes were investigated in carbapenem-resistant isolates using PCR.

DETAILED DESCRIPTION:
Patients with P. mirabilis growth in blood culture who met the study criteria were divided into two groups as carbapenem susceptible and resistant according to carbapenem antibiogram results. Patients with carbapenem-resistant P. mirabilis (CRPM) growth in blood culture were included in the case group and patients with carbapenem- susceptible P. mirabilis (CSPM) growth in blood culture were included in the control group.

Demographic characteristics of the patients, concomitant chronic diseases, Charlson comorbidity index (CCI), hospital and intensive care unit (ICU) hospitalization and number of days in the last year, history and type of invasive intervention in the last three months (surgical-invasive), history of antibiotic use in the last three months and types of antibiotics used (Penicillin, cephalosporin, quinolone, carbapenem, tigecycline, colistin, aminoglycoside), hospitalization unit, total length of hospitalization, sample collection unit, growth result and antibiogram, clinical and laboratory data of the day of growth, sepsis and septic shock evaluated according to systemic inflammatory response syndrome (SIRS) criteria, 30-day mortality and patient outcome information were recorded.

Carbapenemase-producing gene regions were investigated by Polymerase Chain Reaction (PCR) in accessible samples of patients with carbapenem-resistant P. mirabilis growth in blood cultures.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients aged 18 years and older
* P. mirabilis growth in blood cultures

Exclusion Criteria:

* Samples taken in emergency departments, outpatient clinics, day treatment units
* Recurrent growths of the same patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: . Inpatients aged 18 years and older with P. mirabilis growth in blood cultures were included in the study, while samples taken in emergency departments, outpatient clinics, day treatment units and recurrent growths of the same patient were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Carbapenem Use | 1 year
  number of patients using carbapenem before P. mirabilis growth in blood cultures
Intensive Care Units | 1 year
  number of patients admission in ıntensive care units before P. mirabilis growth in blood cultures
Mortality | 30 days
  number of patients who died
Length of hospital stay | 1 year
  Length of hospital stay days
Presence of chronic disease | 1 year
  number of patients with chronic disease

CONTACTS AND LOCATIONS:
Overall Officials: Çağlar IRMAK, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No